CLINICAL TRIAL: NCT03979040
Title: A Comparison of Group Transdiagnostic Behavior Therapy (G-TBT) to Disorder-Specific Group Psychotherapies in the Recovery of Veterans With PTSD, Major Depression and Related Conditions
Brief Title: Comparing Group Therapies for Veterans With Depression and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2910-R
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder; Posttraumatic Stress Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Transdiagnostic Behavior Therapy (Experimental): TBT was developed to address transdiagnostic avoidance via the use of four different types of exposure techniques (situational/in-vivo, physical/interoceptive, thought/imaginal, and [positive] emotional/behavioral activation). From the transdiagnostic avoidance perspective, the four exposure practices are matched to the type(s) of avoidance experienced by patients based upon their cluster of symptoms/disorders. Per protocol, the first six sessions of TBT are designed to educate on, prepare for, and practice the four different types of exposure techniques. The next five sessions are focused on practicing and refining exposure practices as participants work through their lists of avoided situations/sensation/thoughts. The final session reviews treatment progress and relapse prevention strategies.
  Interventions: Behavioral: Group Transdiagnostic Behavior Therapy
- Group Disorder-Specific Therapy (G-DSTs) (Active Comparator): To provide an evidence-based comparison for the G-TBT condition, G-DSTs will be used that are matched to the participant's principal diagnosis. G-DSTs will include groups for the most common principal diagnoses that have VA-approved protocols and training programs, including PTSD (Cognitive Processing Therapy for PTSD) and Major Depressive Disorder (CBT-Depression). Each of these G-DSTs have published manuals for administration and have received extensive support in the literature.
  Interventions: Behavioral: Group Disorder-Specific Therapy (G-DSTs)

INTERVENTIONS:
Behavioral: Group Transdiagnostic Behavior Therapy — TBT was developed to address transdiagnostic avoidance via the use of four different types of exposure techniques (situational/in-vivo, physical/interoceptive, thought/imaginal, and [positive] emotional/behavioral activation). From the transdiagnostic avoidance perspective, the four exposure practices are matched to the type(s) of avoidance experienced by patients based upon their cluster of symptoms/disorders. Per protocol, the first six sessions of TBT are designed to educate on, prepare for, and practice the four different types of exposure techniques. The next five sessions are focused on practicing and refining exposure practices as participants work through their lists of avoided situations/sensation/thoughts. The final session reviews treatment progress and relapse prevention strategies.
  Arms: Group Transdiagnostic Behavior Therapy
Behavioral: Group Disorder-Specific Therapy (G-DSTs) — To provide an evidence-based comparison for the G-TBT condition, G-DSTs will be used that are matched to the participant's principal diagnosis. G-DSTs will include groups for the most common principal diagnoses that have VA-approved protocols and training programs, including PTSD (Cognitive Processing Therapy for PTSD) and Depression (CBT-Depression). Each of these G-DSTs have published manuals for administration and have received extensive support in the literature.
  Arms: Group Disorder-Specific Therapy (G-DSTs)

SUMMARY:
Cognitive behavioral therapy (CBT) is a brief, efficient, and effective psychotherapy for individuals with depressive and PTSD. However, CBT is largely underutilized within Veteran Affairs Medical Centers (VAMCs) due to the cost and burden of trainings necessary to deliver the large number of CBT protocols. Transdiagnostic Behavior Therapy (TBT), in contrast, is specifically designed to address numerous distinct disorders within a single protocol. The transdiagnostic approach of TBT has the potential to dramatically improve the accessibility of CBT within VAMCs and therefore improve clinical outcomes of Veterans. The proposed research seeks to evaluate the efficacy of a group version of TBT (G-TBT) by assessing clinical outcomes and quality of life in VAMC patients with major depressive disorder and PTSD throughout the course of treatment and in comparison to two existing group disorder-specific therapies (G-DST), CBT for Depression and Cognitive Processing Therapy for PTSD.

DETAILED DESCRIPTION:
Objective To examine efficacy of G-TBT on improving quality of life, psychological well-being, and social reintegration of Veterans with PTSD, Major Depressive Disorder, and related conditions compared to G-DSTs using a non-inferiority design. Patient satisfaction, access, and predictors of feasibility (attendance and discontinuation) also will be assessed.

Recruitment Strategy Veterans will be recruited through the Primary Care - Mental Health Integration, General Outpatient Mental Health, and CBT Clinic programs at the Charleston VAMC. Within these programs, all Veterans reporting symptoms of depression and anxiety meet with a mental health staff member to complete a clinical interview and self-report measures. If Veterans endorse symptoms consistent with a depressive/anxiety disorder, interest in participating in research will be assessed and, if agreeable, the Veteran will be referred to project staff. A study-specific intake appointment will be completed with the project staff to assess inclusion/exclusion criteria (with a targeted sample of 326 VAMC patients), including a semi-structured clinical interview and self-report questionnaires focused on quality of life, social integration, and psychiatric symptoms (described later). Participants who meet inclusion/exclusion criteria will be randomized into a study condition, and will be assigned to a project therapist. Because most VAMC patients who meet study criteria likely will present with multiple depressive/anxiety disorders, principal diagnosis, or the most impairing of the diagnosable disorders, will be used to select patients for participation and inform randomization. Principal diagnosis will be determined via diagnostic severity scores in the Anxiety Disorders Interview Schedule-5. To balance diagnoses across the two conditions, a stratified random assignment based on principal diagnosis will be used (Major Depressive Disorder and PTSD).

Procedures Eligible VAMC patients will be randomized into one of two treatment conditions: G-TBT or G-DSTs. Both treatment conditions will include 12 weekly 90-minute group sessions. The general format of sessions will involve: 1) brief check-in; 2) review of materials from previous sessions; 3) review of homework assignments; 4) overview of new materials and in-session exercises; and 5) assignment of homework for next session. Attendance and homework completion will be recorded.

Treatment groups (G-TBT, Group CBT-Depression, Group Cognitive Processing Therapy for PTSD) will require at least 6 participants and maximum of 12 participants to begin. Upon randomization, participants will be notified of the group assignment and expected wait period for the group to begin. Wait periods (in days) will be recorded as an indicator of access to treatment across groups.

Randomization Procedures Participants will be randomly assigned (1:1) to one of the two study arms (n = 104 per arm) using a permuted block randomization procedure. Randomization will be stratified by principal diagnostic group (or most impairing disorder between Major Depressive Disorder and PTSD if both disorders are present, based upon disorder-specific interference and distress severity scores) and block size will be varied to minimize the likelihood of unmasking. If both disorders evidence identical severity scores (highly unlikely), participants will be asked which of the two disorders is more impairing/significant for randomization purposes. After determining eligibility and completing consent and baseline assessment materials, enrolled participants will be assigned to treatment conditions by the Research Coordinator/Therapist using a computer-generated randomization scheme. Once a participant is randomized, they will be included in the intent-to-treat analysis. Randomization will occur at the participant level.

Group Transdiagnostic Behavior Therapy TBT was developed as a streamlined protocol to address transdiagnostic avoidance via the use of four different types of exposure techniques (situational/in-vivo, physical/interoceptive, thought/imaginal, and [positive] emotional/behavioral activation). From the transdiagnostic avoidance perspective, the four exposure practices are matched to the type(s) of avoidance experienced by patients based upon their cluster of symptoms/disorders. Per protocol, the first six sessions of TBT are designed to educate on, prepare for, and practice the four different types of exposure techniques. The next five sessions are focused on practicing and refining exposure practices as participants work through their lists of avoided situations/sensation/thoughts. The final session reviews treatment progress and relapse prevention strategies.

G-DSTs Control Condition Matching and Assignment To provide an evidence-based comparison for the G-TBT condition, G-DSTs will be used that are matched to the participant's principal diagnosis. G-DSTs will include groups for the most common principal diagnoses that have VA-approved protocols and training programs, including PTSD (Cognitive Processing Therapy for PTSD) and Major Depressive Disorder (CBT-Depression). Each of these G-DSTs have published manuals for administration and have received extensive support in the literature. Participants randomized to a G-DST group will be matched to the G-DST based on the principal diagnosis determined via the diagnostic interview.

ELIGIBILITY:
Inclusion Criteria:

* participants must be clearly competent to provide informed consent for research participation;
* participants must meet Diagnostic and Statistical Manual-5 diagnostic criteria for a principal diagnosis of a major depressive disorder or posttraumatic stress disorder
* participant must be a Veteran enrolled at Veterans Affairs Medical center within the Charleston VAMC catchment area

Exclusion Criteria:

* recent history (< 2 months) of psychiatric hospitalization or a suicide attempt as documented in their medical record or reported during clinical interview
* current diagnosis of substance use disorder as documented in their medical record or reported during clinical interview
* acute, severe illness or medical condition that likely will require hospitalization and/or otherwise interfere with study procedures as documented in their medical record (e.g., active chemotherapy/radiation treatment for cancer, kidney dialysis, oxygen therapy for chronic obstructive pulmonary disease),
* recent start of new psychiatric medication (< 4 weeks)
* diagnosis of traumatic brain injury in their medical record and/or endorsement of screener questionnaire regarding the symptoms of traumatic brain injury modified from the Post-Deployment Health Assessment employed by the Department of Defense
* diagnosis of schizophrenia, psychotic symptoms, personality disorder, and/or bipolar disorder as documented in their medical record or reported during clinical interview
* VAMC patients excluded due to these factors will be reconsidered for participation once the condition related to their exclusion is resolved or stabilized
* Ineligible VAMC patients will be referred for non-study-related treatments within mental health at the Ralph H. Johnson VA Medical Center

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Gros, PhD MA BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon consultation with the local VA Research & Development Committee and university-affiliated institutional review board committees after publication of primary research questions, the de-identified database will be made available to the public via the publishing journal's website (where applicable) as well as on (yet to be determined/selected) research community websites designed for the sharing of scientific findings and data.
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication of the primary outcome papers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 294 participants completed the intake procedures and consent documentation. Of the 294, 243 participants met study inclusion/exclusion criteria and were enrolled and randomized to study condition
Groups:
- Group Transdiagnostic Behavior Therapy: TBT was developed to address transdiagnostic avoidance via four exposure practices are matched to the type(s) of avoidance experienced by patients based upon their cluster of symptoms/disorders. Per protocol, the first six sessions of TBT are designed to educate on, prepare for, and practice the four different types of exposure techniques. The next five sessions are focused on practicing and refining exposure practices as participants work through their lists of avoided situations/sensation/thoughts. The final session reviews treatment progress and relapse prevention strategies.
- Group Disorder-Specific Therapy (G-DSTs): To provide an evidence-based comparison for the G-TBT condition, G-DSTs will be used that are matched to the participant's principal diagnosis. G-DSTs included groups for PTSD (Cognitive Processing Therapy for PTSD) and MDD (CBT-Depression). Each of these G-DSTs have published manuals for administration and have received extensive support in the literature.
Period: Overall Study
Arm/Group | Group Transdiagnostic Behavior Therapy | Group Disorder-Specific Therapy (G-DSTs)
Started | 125 | 118
Completed | 69 | 46
Not Completed | 56 | 72
Not completed — Withdrawal by Subject | 24 | 32
Not completed — randomized but never started treatment | 32 | 39
Not completed — withdrawn by study team due to poor fit/lack of efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Transdiagnostic Behavior Therapy | Group Disorder-Specific Therapy (G-DSTs) | Total
Number analyzed (Participants) | 125 | 118 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (12.4) | 45.7 (14.0) | 45.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 32 | 71
  Male | 86 | 86 | 172
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 58 | 57 | 115
  Black, non-Hispanic | 56 | 48 | 104
  Asian American | 1 | 2 | 3
  Hispanic | 6 | 9 | 15
  Native American | 2 | 0 | 2
  Other | 2 | 2 | 4
Depression Anxiety Stress Scales - Depression (DASS-D) [Mean (Standard Deviation); unit: units on a scale] — The DASS-Depression is a 7-item measure designed to assess dysphoric mood. Items are rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), and summed to compute the total scale that ranges from 0 to 21. Higher scores are indicative of greater symptom severity. The factor structure, reliability, and validity of the subscales have been supported in the literature. Population: A number of participants were randomized based on completing consent documents and diagnostic assessment (inclusion/exclusion criteria), but failed to mail in their baseline symptom measures.
  units on a scale
    number analyzed (Participants) | 81 | 78 | 159
    (all) | 10.8 (5.3) | 12.0 (5.5) | 11.4 (5.4)
PTSD Checklist for DSM-5 (PCL) [Mean (Standard Deviation); unit: units on a scale] — The PCL-5 is a 20-item self-report measure that assesses DSM-5 criteria PTSD symptoms. Items are rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (extremely), and summed to compute the total scale that ranges from 0 to 80. Higher scores are indicative of greater symptom severity. Previous versions of the PCL have been shown to have excellent internal consistency and excellent test-retest reliability in veterans. In addition, the PCL-5 has been incorporated into standard assessment for PTSD at the VA. Population: A number of participants were randomized based on completing consent documents and diagnostic assessment (inclusion/exclusion criteria), but failed to mail in their baseline symptom measures.
  units on a scale
    number analyzed (Participants) | 80 | 78 | 158
    (all) | 43.7 (17.2) | 46.2 (14.2) | 44.9 (15.8)
Illness Intrusiveness Ratings Scale (IIRS) [Mean (Standard Deviation); unit: units on a scale] — The IIRS is a 13-item questionnaire that assesses the extent to which a disease interferes with important domains of life, including health, diet, work, and several others. Each item is rated on a 7-point Likert scale, ranging from 1 (not very much) to 7 (very much). Items are summed to create the total score (ranging from 1 to 91), with higher scores indicative of greater impairment. The IIRS has been shown to have high internal consistency in the previous literature. Population: A number of participants were randomized based on completing consent documents and diagnostic assessment (inclusion/exclusion criteria), but failed to mail in their baseline symptom measures.
  units on a scale
    number analyzed (Participants) | 81 | 78 | 159
    (all) | 60.4 (14.6) | 61.4 (16.5) | 60.9 (15.5)

OUTCOME MEASURES:

1. Primary Outcome: Depression Anxiety Stress Scale (DASS-Depression)
Description: The DASS-Depression is a 7-item measure designed to assess dysphoric mood. Items are rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), and summed to compute the total scale that ranges from 0 to 21. Higher scores are indicative of greater symptom severity. The factor structure, reliability, and validity of the subscales have been supported in the literature.
Time Frame: change from baseline to 6-month follow-up
Population: The total number of participants analyzed is inconsistent from the total number of participants reported in the Participant Flow due to missing data - participants failed to return self-report questionnaire packets.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Transdiagnostic Behavior Therapy | Group Disorder-Specific Therapy (G-DSTs)
Number analyzed (Participants) | 51 | 35
units on a scale
  mid-treatment (week 6) | 10.6 (5.8) | 11.0 (5.9)
  post-treatment (week 12): number analyzed (Participants) | 41 | 29
  post-treatment (week 12) | 8.8 (6.1) | 8.1 (5.9)
  follow-up (6 months post-treatment): number analyzed (Participants) | 36 | 29
  follow-up (6 months post-treatment) | 8.5 (6.9) | 9.9 (6.4)
Statistical Analysis 1: Comparison: Group Transdiagnostic Behavior Therapy vs Group Disorder-Specific Therapy (G-DSTs); Test type: Non-Inferiority — A non-inferiority margin of -.5 was set for outcome analysis with a one-sided alpha of .025; p = .025, Sign test — P value = .025 (one-sided) and sign test below; Mean Difference (Net) = -.5

2. Primary Outcome: Illness Intrusiveness Ratings Scale (IIRS)
Description: The IIRS is a 13-item questionnaire that assesses the extent to which a disease interferes with important domains of life, including health, diet, work, and several others. Each item is rated on a 7-point Likert scale, ranging from 1 (not very much) to 7 (very much). Items are summed to create the total score (ranging from 1 to 91), with higher scores indicative of greater impairment. The IIRS has been shown to have high internal consistency in the previous literature.
Time Frame: change from baseline to 6-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Transdiagnostic Behavior Therapy | Group Disorder-Specific Therapy (G-DSTs)
Number analyzed (Participants) | 51 | 35
units on a scale
  mid-treatment (week 6) | 62.6 (17.8) | 59.3 (15.5)
  post-treatment (week 12): number analyzed (Participants) | 41 | 29
  post-treatment (week 12) | 59.0 (18.1) | 52 (19.2)
  follow-up (6-months post-treatment): number analyzed (Participants) | 36 | 29
  follow-up (6-months post-treatment) | 53.8 (23.8) | 52.9 (22.7)
Statistical Analysis 1: Comparison: Group Transdiagnostic Behavior Therapy vs Group Disorder-Specific Therapy (G-DSTs); Test type: Non-Inferiority — A non-inferiority margin of -.5 was set for outcome analysis with a one-sided alpha of .025; p = .025, Sign test; Mean Difference (Net) = -.5

3. Primary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: The PCL-5 is a 20-item self-report measure that assesses DSM-5 criteria PTSD symptoms. Items are rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (extremely), and summed to compute the total scale that ranges from 0 to 80. Higher scores are indicative of greater symptom severity. Previous versions of the PCL have been shown to have excellent internal consistency and excellent test-retest reliability in veterans. In addition, the PCL-5 has been incorporated into standard assessment for PTSD at the VA.
Time Frame: change from baseline to 6-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Transdiagnostic Behavior Therapy | Group Disorder-Specific Therapy (G-DSTs)
Number analyzed (Participants) | 50 | 34
units on a scale
  mid-treatment (week 6) | 43.4 (19) | 40.0 (15.5)
  post-treatment (week 12): number analyzed (Participants) | 41 | 29
  post-treatment (week 12) | 40.3 (18.3) | 33.9 (18.5)
  follow-up (6-month post-treatment): number analyzed (Participants) | 35 | 29
  follow-up (6-month post-treatment) | 36.9 (20.5) | 35.9 (20.6)
Statistical Analysis 1: Comparison: Group Transdiagnostic Behavior Therapy vs Group Disorder-Specific Therapy (G-DSTs); Test type: Non-Inferiority — A non-inferiority margin of -.5 was set for outcome analysis with a one-sided alpha of .025; p = .025, Sign test; Mean Difference (Net) = -.5

ADVERSE EVENTS:
Time Frame: Unexpected/serious adverse events were monitored throughout the duration of the active treatment phase of the study for each participant (e.g., baseline to 6-month follow-up assessment, or an average of 10 months).
Description: Due to the nature of the study treatment (group psychotherapy), the study focused on unexpected serious adverse events.
Arm/Group | Group Transdiagnostic Behavior Therapy | Group Disorder-Specific Therapy (G-DSTs)
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/118
Other Adverse Events (participants affected / at risk) | 0/125 | 0/118

LIMITATIONS AND CAVEATS:
Recruitment was set to begin in Spring 2020. The COVID pandemic resulted in significant delays, as well as in changes in the methods of the study (e.g., shifted to telehealth). These two changes likely contributed in the higher-than-expected treatment discontinuation (group psychotherapy via telehealth) and missing data (traditional mail delivery-return of questionnaires). The target sample was increased to adjust for the missing data based on updated power analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT03979040/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT03979040/ICF_000.pdf